CLINICAL TRIAL: NCT02746094
Title: Low Frequency Shock Wave Therapy for Improving Post-prostatectomy Erectile Dysfunction: a Prospective Pilot Study
Acronym: ProstaChoc 1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change strategy
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Direx Systems GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2016/SD-01
Record Dates: First submitted 2016-04-13; First posted 2016-04-21 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study population (Experimental): The study population is comprised of adult men less than 80 years of age who are consulting for ED lasting for over 6 months following a prostatectomy that took place 18 to 60 months ago. The patients are currently in a stable relationship that has been going on for at least 3 months, have an IIEF-EF score between 6 and 25, and have at least a natural tumescence during sexual stimulation (EHS score ≥ 1).
  Intervention: 8 bi-weekly LIESWT sessions
  Interventions: Device: 8 bi-weekly LIESWT sessions

INTERVENTIONS:
Device: 8 bi-weekly LIESWT sessions — LIESWT = Low-Intensity Extracorporeal Shock Wave Therapy
  The treatment protocol consists of eight bi-weekly treatment sessions (weeks 0 ot 4). During each session 3600 shocks at 0.09 mJ/mm are applied. Shocks are applied to the penis shaft at the right corpus cavernosum and the left corpus cavernosum, and at the crura at the right crus and the left crus. 900 shocks are administered to each area. The treatment areas are the same for each session, so that at the end of the full treatment (8 sessions) each area will have received 7200 shocks at 0.09 mJ/mm.
  In general, the patient is placed on an examination table. A series of focused shockwaves produced by the electromagnetic transducer are coupled to a patient's penile shaft and crura and are made to converge along the penis/crura volume. The operator controls treatment parameters including shockwave intensity and shockwave rate.
  mJ = millijoule.
  Other Names: RENOVA device

SUMMARY:
The primary objective of this study is to evaluate changes in erectile function (EF) before versus after 8 bi-weekly treatments of Low-Intensity Extracorporeal Shock Wave Therapy (LIESWT) via IIEF-EF (the Erectile Function domain of the International Index of Erectile Function) scores.

DETAILED DESCRIPTION:
The secondary objectives of this study are to evaluate changes in the following elements before versus after 8 bi-weekly treatments of LIESWT:

A. EF categorical improvement.

B. Other validated measures of EF (SEP2 (question 2 of the sexual encounter profile), SEP3 (question 3 of the sexual encounter profile), GAQ (Global Assessment Question), EHS (Erection Hardness Score)), and the remaining domains of the IIEF score (orgasmic function, sexual desire, intercourse satisfaction, overall satisfaction), as well as the total IIEF score.

C. Harms/Safety: To evaluate treatment tolerance and potential adverse events.

ELIGIBILITY:
Inclusion Criteria:

* The patient has given his informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is a man at least 18 years old and less than 80 years old
* The patient has been in a stable, sexual relationship with only one other person for at least the past three months
* The patient is consulting for erectile dysfunction lasting for over 6 months
* The patient had a prostatectomy 18 to 60 months ago
* The patient has an erectile function domain score on the International Index of Erectile Function questionnaire between 6 and 25
* The patient has at least a natural tumescence during sexual stimulation (erection hardness score ≥ 1)
* The patient has not had phosphodiesterase type 5 inhibitor treatment for the month preceding inclusion
* The patient is available for 8 months of follow-up and agrees to participate in all study visits

Exclusion Criteria:

* The patient is participating in another interventional study, or has participated in another interventional study within the past 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or is an adult under guardianship
* It is impossible to correctly inform the patient, or the patient refuses to sign the consent
* Complete anerection
* Untreated testosterone deficiency
* Neurological disease
* Psychiatric disease
* Anatomical malformation of the penis
* Chronic haematological pathology with significant clinical impact
* Oral or injectable antiandrogen treatment
* The patient is taking blood thinners and has an international normalized ratio > 3
* History of erectile dysfunction before the prostatectomy

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
The difference in the rate of change for the IIEF-EF score before and after treatment sessions (change per two-month period). | rate of change between -8 and 0 weeks versus rate of change between 0 and 8 weeks
  IIEF-EF = the erectile function domain of the International Index of Erectile Function

SECONDARY OUTCOMES:
The change in the number of patients with improvement in erectile function (EF) over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | -8 to 0 weeks versus 0 to 8 weeks
  Improvement in EF is defined as a >2 point increase in the IIEF-EF score from baseline for mild erectile dysfunction (ED), >5 points for moderate ED and >7 points for severe ED (Rosen et al. 2011).
The change in the number of patients with improvement in erectile function (EF) over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | -8 to 0 weeks versus 0 to 16 weeks
  Improvement in EF is defined as a >2 point increase in the IIEF-EF score from baseline for mild erectile dysfunction (ED), >5 points for moderate ED and >7 points for severe ED (Rosen et al. 2011).
The change in the number of patients with improvement in erectile function (EF) over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | 0 to 8 weeks versus 8 to 16 weeks
  Improvement in EF is defined as a >2 point increase in the IIEF-EF score from baseline for mild erectile dysfunction (ED), >5 points for moderate ED and >7 points for severe ED (Rosen et al. 2011).
The change in the number of patients responding yes to question 2 of the Sexual Encounter Profile over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | -8 to 0 weeks versus 0 to 8 weeks
  Were you able to insert your penis into your partner's vagina? (yes/no)
The change in the number of patients responding yes to question 2 of the Sexual Encounter Profile over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | -8 to 0 weeks versus 0 to 16 weeks
  Were you able to insert your penis into your partner's vagina? (yes/no)
The change in the number of patients responding yes to question 2 of the Sexual Encounter Profile over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | 0 to 8 weeks versus 8 to 16 weeks
  Were you able to insert your penis into your partner's vagina? (yes/no)
The change in the number of patients responding yes to question 3 of the Sexual Encounter Profile over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | -8 to 0 weeks versus 0 to 8 weeks
  Did your erection last long enough for you to have successful intercourse? (yes/no)
The change in the number of patients responding yes to question 3 of the Sexual Encounter Profile over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | -8 to 0 weeks versus 0 to 16 weeks
  Did your erection last long enough for you to have successful intercourse? (yes/no)
The change in the number of patients responding yes to question 3 of the Sexual Encounter Profile over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | 0 to 8 weeks versus 8 to 16 weeks
  Did your erection last long enough for you to have successful intercourse? (yes/no)
The change in the number of patients responding yes to the Global Assessment Question (yes/no) over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | -8 to 0 weeks versus 0 to 8 weeks
  Has the treatment you have been taking improved your erectile function? (yes/no)
The change in the number of patients responding yes to the Global Assessment Question (yes/no) over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | -8 to 0 weeks versus 0 to 16 weeks
  Has the treatment you have been taking improved your erectile function? (yes/no)
The change in the number of patients responding yes to the Global Assessment Question (yes/no) over a period of observation before the treatment sessions versus a period of observation after the start of treatment sessions. | 0 to 8 weeks versus 8 to 16 weeks
  Has the treatment you have been taking improved your erectile function? (yes/no)
The difference in the rate of change for the total IIEF score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 8 weeks
The difference in the rate of change for the total IIEF score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 16 weeks
The difference in the rate of change for the IIEF erectile function subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 8 weeks
The difference in the rate of change for the IIEF erectile function subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 16 weeks
The difference in the rate of change for the IIEF sexual satisfaction subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 8 weeks
The difference in the rate of change for the IIEF sexual satisfaction subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 16 weeks
The difference in the rate of change for the IIEF orgasmic function subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 8 weeks
The difference in the rate of change for the IIEF orgasmic function subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 16 weeks
The difference in the rate of change for the IIEF sexual desire subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 8 weeks
The difference in the rate of change for the IIEF sexual desire subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 16 weeks
The difference in the rate of change for the IIEF overall satisfaction subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 8 weeks
The difference in the rate of change for the IIEF overall satisfaction subdomain score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 16 weeks
The difference in the rate of change for the EHS Score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 8 weeks
The difference in the rate of change for the EHS Score before and after treatment sessions (change per two-month period) | rate of change between -8 and 0 weeks versus rate of change between 0 and 16 weeks
Visual analog scale for pain during treatment (score from 0 to 10) | Week 1, Monday or Tuesday
Visual analog scale for pain during treatment (score from 0 to 10) | Week 1, Thursday or Friday
Visual analog scale for pain during treatment (score from 0 to 10) | Week 2, Monday or Tuesday
Visual analog scale for pain during treatment (score from 0 to 10) | Week 2, Thursday or Friday
Visual analog scale for pain during treatment (score from 0 to 10) | Week 3, Monday or Tuesday
Visual analog scale for pain during treatment (score from 0 to 10) | Week 3, Thursday or Friday
Visual analog scale for pain during treatment (score from 0 to 10) | Week 4, Monday or Tuesday
Visual analog scale for pain during treatment (score from 0 to 10) | Week 4, Thursday or Friday
The presence/absence any other complications that might occur (almost none are cited in the literature) | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Droupy, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Background] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209